CLINICAL TRIAL: NCT00711997
Title: Phase 1/2a, Dose-Escalation, Safety, Pharmacokinetic, and Preliminary Efficacy Study of Intratumoral Administration of DTA-H19 in Patients With Unresectable Pancreatic Cancer
Brief Title: Phase 1/2a DTA-H19 in Patients With Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-07-05
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Neoplasms
Keywords: H19 gene, plasmid, diphtheria toxin, pancreatic cancer; inodiftagene vixteplasmid; BC-819
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BC-819 (Experimental): Intratumoral administration of BC-819
  Interventions: Biological: DTA-H19

INTERVENTIONS:
Biological: DTA-H19 — Cohort #1: 4 mg DTA-H19 intratumorally 2 times per week for 2 weeks Cohort #2: 8 mg DTA-H19 intratumorally 2 times per week for 2 weeks
  Other Names: BC-819

SUMMARY:
This study is designed to assess the safety, tolerability, pharmacokinetics (PK) and preliminary efficacy of DTA-H19 administered intratumorally in patients with unresectable, locally advanced pancreatic cancer.

Primary Objective: The primary objective is to determine the maximum tolerated dose (MTD) of intratumoral DTA-H19 and identify any dose limiting toxicities (DLTs).

Secondary objectives include determining the adverse events (AEs) profile, effects on clinical laboratory analytes, vital signs, PK, tumor response, and possible tumor resectability after 4 intratumoral administrations of DTA-H19.

DETAILED DESCRIPTION:
DTA-H19, is a doubled stranded DNA plasmid that carries the gene for the diphtheria toxn A (DT-A) chain under the regulation of the H19 promoter sequence. This is a Patient-Oriented, Targeted Therapy as DT-A chain expression is triggered by the presence of H19 transcription factors that are upregulated in tumor cells. The selective initiation of toxin expression results in selective tumor cell destruction via inhibition of protein synthesis in the tumor cell, enabling highly targeted cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and be between the ages of 18 and 79, inclusive.
* Have unresectable, locally advanced adenocarcinoma of the pancreas proven by biopsy or cytology (defined as direct extension to the superior mesenteric artery and/or celiac axis with loss of a clear plane between tumor and these arterial structures, or loss of patent superior mesenteric-portal vein confluence). Patients who have been surgically explored and deemed unresectable on that basis are eligible, provided other entry criteria are met. Patients having potentially resectable regional lymph node involvement may be included.
* Have a target tumor ≤ 6 cm in diameter that is accessible for intratumoral administration by PTA or EUS guidance as determined by the radiologist/gastroenterologist performing the PTA/EUS injection.
* Have a Karnofsky performance status of ≥ 70%.
* Have a life expectancy of >= 3 months.
* If female and of child-bearing potential, have a negative serum pregnancy test during screening.
* Agree to use of a barrier method of contraception if sexually active (both men and women) from the time of administration of the first treatment and for at least 8 weeks after treatment.
* Have serum creatinine < 2.0 mg/dL, AST and ALT >= 2.5 x ULN, PT, PPT, and PT/INR within normal limits, absolute neutrophil count (ANC) > 1,500 x 103 cells/mL, platelets ≥ 100,000/mL, and hemoglobin >= 10 mg/dL.
* Have a biopsy specimen that is positive for H19 expression (grade 2 or greater staining determined by a pathologist).
* Have screening procedures completed within 4 weeks of starting treatment.
* No other malignancy present that would interfere with the current intervention.
* Commit to refrain from any concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol, therefore any standard treatment should be postponed while on study.
* Have measurable disease.

Exclusion Criteria:

* Have distant metastatic spread (such as liver or lung metastases), peritoneal spread or malignant ascites.
* Have prior radiation therapy for pancreatic cancer or radiation to the area of the target tumor field.
* Endocrine tumors or lymphoma of the pancreas.
* Have clinically significant pancreatitis within 12 weeks of treatment.
* If female, be breast feeding.
* Have a medical condition contraindicated for both percutaneous- and endoscopic- guided delivery or any intercurrent medical illness or other medical condition that would in the judgment of the investigator compromise patient safety or the objectives of the study.
* Have a history of coagulopathy.
* Have participated in any therapeutic research study within the last 4 weeks.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Czerniak, MD, Principal Investigator — The Chaim Sheba Medical Center; Nader Hanna, MD, FACS, Principal Investigator — University of Maryland; Fred Konikoff, MD, Principal Investigator — Meir Medical Center; Ayala Hubert, MD, Principal Investigator — Hadassah University Hospital
Locations (4):
- University of Maryland Medical Center, Baltimore, Maryland, United States
- Israel (3):
  - Hadassah University Hospital, Jerusalem
  - Meir Hospital, Kfar Saba
  - The Chaim Sheba Medical Center, Tel Litwinsky

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 26 Oct 2009 Last subject completed: 7 Oct 2010 at 4 medical centers in Israel an 1 in US
Pre-assignment Details: Of the 16 patients screened, 7 were screening failures due to metastatic disease
Groups:
- BC-819 4 mg: Each cohort of 3 to 6 subjects received 2 weeks of twice weekly intratumoral injections of BC-819. Intratumoral injections were performed using PTA- or EUS-guided administrations of BC-819. For each treatment, this cohort received a single injection of 1 mL of 4 mg/mL for a total of 4 mg of BC-819 per injection.
- BC-819 8 mg: Each cohort of 3 to 6 subjects received 2 weeks of twice weekly intratumoral injections of BC-819. Intratumoral injections were performed using PTA- or EUS-guided administrations of BC-819. For each treatment, this cohort received a single injection of 2 mL of 4 mg/mL for a total of 8 mg of BC-819.
Period: Overall Study
Arm/Group | BC-819 4 mg | BC-819 8 mg
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BC-819 4 mg | BC-819 8 mg | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (18.3) | 60 (10) | 62 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 0 | 1 | 1
  Israel | 3 | 5 | 8

OUTCOME MEASURES:

1. Secondary Outcome: Tumor Response
Description: Tumor response and progression were defined in accordance with RECIST v. 1.0 and assessed by radiological examination 2 weeks after the end of treatment
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | BC-819 4 mg | BC-819 8 mg
Number analyzed (Participants) | 3 | 6
participants
  Stable disease | 1 | 4
  Progressive disease | 2 | 2

2. Secondary Outcome: Tumor Resectability
Description: The number of subjects in each cohort whose tumor was resectable at the end of the study was to be presented for the ITT and the per-protocol population.
Time Frame: 5 to 6 weeks
Measure: Number; unit: participants
Arm/Group | BC-819 4 mg | BC-819 8 mg
Number analyzed (Participants) | 3 | 6
participants | 0 | 1

3. Primary Outcome: Maximal Tolerated Dose (MTD) & Dose Limiting Toxicity (DLT) of Intratumoral Injections of BC-819
Description: If 2 patients in any cohort experience DLTs, then the next lower dose will be considered the MTD if there is a lower dose cohort. A DLT is defined as grade 3 or greater toxicity judged to be at least possibly related to the investigational products.
Time Frame: Week 4
Population: All participants had to receive all 4 scheduled treatments and completed the Week 4 assessment
Measure: Number; unit: participants
Groups:
- BC-819 4 mg: 1 mL of 4 mg/mL for a total of 4 mg of BC-819 per injection for 2 weeks of twice weekly intratumoral BC-819. Intratumoral injections were performed using CT-guided PTA or EUS of BC-819.
- BC-819 8 mg: 2 mL of 4 mg/mL for a total of 4 mg of BC-819 per injection for 2 weeks of twice weekly intratumoral BC-819. Intratumoral injections were performed using CT-guided PTA or EUS of BC-819.
Arm/Group | BC-819 4 mg | BC-819 8 mg
Number analyzed (Participants) | 3 | 6
participants | 0 | 1

ADVERSE EVENTS:
Groups:
- BC-819 4 mg: 1 mL of 4 mg/mL for a total of 4 mg of BC-819 per injection for 2 weeks of twice weekly intratumoral BC-819.
- BC-819 8 mg: 2 mL of 4 mg/mL for a total of 8 mg of BC-819 per injection for 2 weeks of twice weekly intratumoral BC-819.
Arm/Group | BC-819 4 mg | BC-819 8 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BC-819 4 mg (N=3) | BC-819 8 mg (N=6)
Abdominal pain & Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lab abnormalities (Investigations) | 3 (7) | 6 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
General disorders (General disorders) | 0 (0) | 1 (4)
Hyperglycemia & hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vasovagal syncope (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No